CLINICAL TRIAL: NCT05872386
Title: "Bupe by the Book": Developing and Testing a Tele-Buprenorphine Intervention in Public Libraries With Unstably Housed Persons With Opioid Use Disorder
Brief Title: "Bupe by the Book": A Tele-Buprenorphine Clinical Trial in Public Libraries With Unstably Housed Persons With Opioid Use Disorder
Acronym: BBB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other)
Responsible Party: Principal Investigator, Lianne Urada, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BBB
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Telehealth at the Library; Control Group
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: We will conduct a 12-week pilot 2-arm randomized controlled trial (RCT) (n=40-60). Research staff will recruit library patrons and randomize them to weekly telehealth at the library or in-person clinic control arms across two participating libraries in San Diego.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth (Experimental): Intervention arm
  Interventions: Behavioral: Buprenorphine uptake/retention via Telehealth
- Treatment as Usual (Experimental): Treatment as usual (in-person at clinic)
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Buprenorphine uptake/retention via Telehealth — Bupe by the Book (BBB) randomly assigns unstably housed library patrons with opioid use disorder to a telehealth to receive buprenorphine (aka, Suboxone) treatment from Father Joe's Villages Health Center.
  Arms: Telehealth
Behavioral: Control group — unstably housed library patrons with opioid disorder are assigned randomly to a treatment as usual control group (in-person at the clinic)
  Arms: Treatment as Usual

SUMMARY:
Public libraries nationwide are facing an on-premise opioid overdose crisis. Many persons with opioid use disorder (OUD) remained unhoused and profoundly hard to reach. This study innovatively develops and tests a telemedicine intervention delivered through public libraries to increase unstably housed individuals' access to bupe treatment that would prevent overdoses from occurring in the first place. The investigators will conduct a 12-week pilot 2-arm randomized controlled trial (RCT) (n=40). Research staff will recruit library patrons and randomize them to weekly telehealth at the library or in-person clinic control arms across two participating libraries in San Diego.

DETAILED DESCRIPTION:
Libraries have become places of refuge for unstably housed individuals with OUD. "Two overdoses a day" occurred just outside the library, according to focus group participants in the investigator's 2019 study on Homelessness in Public Spaces: An Assessment at the San Diego Central Library. Libraries have already taken extraordinary measures to help unstably housed patrons with OUD. The San Diego Central Library trained security staff to carry Narcan to save patrons who overdose in their bathrooms. To deal with daily patron mental health crises, libraries now have social workers, nurses, and peer homeless outreach staff on-site. Buprenorphine "bupe" is a highly effective medical treatment for OUD. However, the investigator's preliminary work shows that unstably housed persons with OUD at libraries perceive lack of bupe access due to transportation and medical coverage issues as barriers to treatment.

"Bupe by the Book" (BBB), in collaboration with the investigators' established local partners, San Diego Public Libraries and Father Joe's Village Health Center (FJV), will innovatively adapt FJV's already successful same-day, free tele-bupe treatment to library settings where OUD patrons are already. BBB will be a groundbreaking 12-week intervention that leverages the library's resources to facilitate low-barrier tele-bupe care via local clinic providers without requiring access to a clinic. By testing BBB uptake and retention in libraries, this study will inform how unstably housed persons and others can receive bupe care in innovative ways with minimal clinical/non-clinical requirements (e.g., low-barrier induction), changing the landscape radically for implementing bupe.

Using a mixed methods approach, the study combines qualitative and quantitative methodologies to address three specific aims:

1. Develop "Bupe by the Book" (BBB) within TAM: Through formative research using intervention mapping, the investigators will conduct a series of 8 focus groups across 4 libraries to: a) assess perceptions of key stakeholders such as local residents, businesses, library staff/security, outreach workers, tele-bupe providers, and unstably housed persons with OUD about BBB's potential, b) develop a feasible plan with stakeholder input, and c) identify facilitators and modifiable barriers to implementation.
2. Determine the feasibility of BBB: Estimate the expected level of treatment uptake and adherence. The investigators will conduct a 12-week pilot 2-arm randomized controlled trial (RCT) (n=40). Research staff will recruit library patrons and randomize them to weekly telehealth at the library or in-person clinic control arms across two participating libraries in San Diego. A health provider at FJV will then screen participants in person for eligibility for same-day bupe induction. BBB's effects on bupe induction and adherence to prescribed doses will be based on self-reported measures at 1-,2-,4-,8-, 12- weeks follow-ups with study staff, and weekly drug screenings and prescription pickups. The study hypothesizes that the BBB vs. control group, will have higher uptake and longer adherence to treatment.
3. Evaluate the acceptability of BBB: Identify program components that could be improved to enhance adherence and patient satisfaction. Research staff will conduct structured interviews with BBB patients, health providers, and library staff to gain insight into the patients' experiences after receiving BBB.

In line with NIDA's 2020 Strategic Plan (Objective 3.4. Develop and test strategies for effectively and sustainably implementing evidence-based treatments), the proposed study addresses long-standing barriers to bupe uptake/adherence. By utilizing multiple library sites, the investigators will render tele-bupe reproducible for other libraries nationwide facing opioid overdoses. This work will pave the foundation for a larger RCT in a subsequent R01 to evaluate the efficacy of utilizing public settings to treat substance use disorders and reduce opioid-related deaths.

ELIGIBILITY:
Inclusion Criteria:

* All participants interested in OUD treatment will be eligible for study screening regardless of OUD and treatment history. However, they cannot already be on bupe with an active medical prescriber unless they can no longer stay with that provider. We will accommodate participants with disabilities. The FJV medical provider will determine if bupe is appropriate for the individual and able to proceed in BBB.

Exclusion Criteria:

* Persons with comorbidities or polysubstance use that needs a different level or type of care from bupe will not be enrolled in either study arm. Participants ineligible for FJV or the libraries will be ineligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
buprenorphine uptake | within first 2 weeks
  participants will pick up prescriptions and take them
buprenorphine adherence | 8-12 weeks
  participants will adhere to prescription by taking buprenorphine for > 1 times and ideally for at least 8 weeks

SECONDARY OUTCOMES:
adherence to appointments | 1-12 weeks
  adherence to appointments
telebupe feasibility | 1-12 weeks
  adherence to telehealth
Opioid use/overdose and other substance use | 1,2,4,8,and 12 weeks
  weekly biomarkers (urinary or oral drug and fentanyl screenings/self-tests) and self-report from surveys

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share individual-level data with the internal research team, including partners at Father Joe's Villages Health Center (FQHC) to obtain their data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: During the study (until June 2024) and after until study closure (approx. 5 years).
Access Criteria: Researchers or data specialists at FJVHC partnering with the BBB researchers.

REFERENCES:
- [Derived] Urada LA, Marienfeld C, Partch M, Garfein RS, Strathdee SA, Nicholls MJ, Weitensteiner A, Zuniga ML, Davidson P, Pitpitan EV. "Bupe by the book": A study protocol for a pilot randomized controlled trial of library-facilitated telehealth to increase buprenorphine treatment among individuals experiencing homelessness. Addict Sci Clin Pract. 2025 Sep 17;20(1):74. doi: 10.1186/s13722-025-00599-2. PMID 40958110
- [Derived] Urada LA, Marienfeld C, Partch M, Garfein RS, Strathdee SA, Nicholls MJ, Weitensteiner A, Zuniga ML, Davidson P, Pitpitan E. "Bupe by the Book": A study protocol for a pilot randomized controlled trial of library-facilitated telehealth to increase buprenorphine treatment among unstably housed individuals. Res Sq [Preprint]. 2024 Nov 25:rs.3.rs-5507141. doi: 10.21203/rs.3.rs-5507141/v1. PMID 39649172